CLINICAL TRIAL: NCT04358211
Title: Convalescent Plasma to Treat and Prevent Pulmonary Complications Associated With COVID-19
Brief Title: Expanded Access to Convalescent Plasma to Treat and Prevent Pulmonary Complications Associated With COVID-19
Status: No longer available | Type: Expanded Access
Sponsor: Nakhle Saba, MD (Other)
Responsible Party: Sponsor-Investigator, Nakhle Saba, MD, Associate Professor of Clinical Medicine, Tulane University School of Medicine
Organization: Tulane University (Other)
Other Study IDs: 2020-595
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Biological: Biological: COVID-19 convalescent plasma — One unit of ABO compatible COVID-19 convalescent plasma

SUMMARY:
I. Study Design: This is a single-arm feasibility study to assess the safety and efficacy of anti-SARS-CoV-2 convalescent plasma (CP) in

1. intubated, mechanically ventilated patients with confirmed COVID-19 pneumonia by chest X-ray or chest CT.
2. hospitalized patients with acute respiratory symptoms between 3 and 7 days after the onset of symptoms, with COVID-19.

II. Study Population:

1. Population 1: Mechanically ventilated intubated COVID-19 patients aged 18 years or older.
2. Population 2: Hospitalized COVID-19 patients aged ≥18 years of age with respiratory symptoms within 3 to 7 days from the beginning of illness.

III. Study Agent:

SARS-CoV-2 convalescent plasma (1-2 units; ~200-400 mL at neutralization antibody titer >1:160.

DETAILED DESCRIPTION:
There are currently no proven safe and efficacious treatment for COVID-19. While most patients recover on their own with basic measures at home, around 20% suffer a more aggressive disease requiring hospitalization, of which 5% necessitating intensive care unit (ICU) admission and potential invasive breathing support. The wide spectrum of COVID 19 also include a significant number of totally asymptomatic patients who are unknowingly spreading the disease. Human convalescent plasma is an option for treatment of COVID-19 and could be rapidly available when there are sufficient numbers of people who have recovered and can donate high titer neutralizing immunoglobulin-containing plasma. This convalescent plasma could be beneficial, not only for severely ill and intubated patients, but also for those with moderate disease early in their disease course to prevent further disease progression and ICU admission.

I. Study Design: This is a single-arm feasibility study to assess the safety and efficacy of anti-SARS-CoV-2 convalescent plasma (CP) in

1. intubated, mechanically ventilated patients with confirmed COVID-19 pneumonia by chest X-ray or chest CT.
2. hospitalized patients with acute respiratory symptoms between 3 and 7 days after the onset of symptoms, with COVID-19.

II. Study Population:

1. Population 1: Mechanically ventilated intubated COVID-19 patients aged 18 years or older.
2. Population 2: Hospitalized COVID-19 patients aged ≥18 years of age with respiratory symptoms within 3 to 7 days from the beginning of illness.

III. Study Duration: April 3, 2020 to December 31, 2022.

IV. Study Agent:

SARS-CoV-2 convalescent plasma (1-2 units; ~200-400 mL at neutralization antibody titer >1:160. (Note this is a moving target as assays develop)). Product will be produced using Blood Bank of New Orleans and safety procedures and procured from patients who have been symptom free for 14 days and screen negative via NP swab or any other test that emerges in the meantime. Doors who have been symptoms free for more than 28 days are eligible to donate without the need of a NP swab. Any emerging FDA guidance will be followed.

ELIGIBILITY:
Inclusion Criteria:

Population 1: Associated Severe Pulmonary Complications

* 18 years or older.
* Hospitalized and intubated in the ICU with COVID-19 respiratory symptoms and confirmation via COVID-19 SARS-CoV-2 RT-PCR testing. Patient or proxy is willing and able to provide written informed consent and comply with all protocol requirements, or requirement for informed consent is WAIVED due to the inability to communicate with the patient and unable to identify legally authorized representative.
* Consents to storage of specimens for future testing, or consent waived.
* The requirements to waive a consent are delineated in 21 CFR 50.23 and will be followed.
* Pregnant and breastfeeding women will not be excluded from the study.

Population 2: Coronavirus Associated Complications in hospitalized patients

* Patients must be 18 years of age or older.
* Hospitalized with COVID-19 respiratory symptoms and confirmation via COVID-19 SARS-CoV-2 RT-PCR testing. Patient is willing and able to provide written informed consent and comply with all protocol requirements.
* Patient agrees to storage of specimens for future testing.

Exclusion Criteria:

Population 1:

* Contraindication to transfusion (severe volume overload, history of anaphylaxis to blood products).
* Severe multi-organ failure with expected life expectancy < 24h as determined by the treating physician.

Population 2:

* Female subjects with positive pregnancy test, breastfeeding, or planning to become pregnant/breastfeed during the study period.
* Receipt of pooled immunoglobulin in past 30 days.
* Contraindication to transfusion or history of prior reactions to transfusion blood products.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Tulane Medical Center, New Orleans, Louisiana, United States

REFERENCES:
- [Result] van Erp EA, Luytjes W, Ferwerda G, van Kasteren PB. Fc-Mediated Antibody Effector Functions During Respiratory Syncytial Virus Infection and Disease. Front Immunol. 2019 Mar 22;10:548. doi: 10.3389/fimmu.2019.00548. eCollection 2019. PMID 30967872
- [Result] Wan Y, Shang J, Sun S, Tai W, Chen J, Geng Q, He L, Chen Y, Wu J, Shi Z, Zhou Y, Du L, Li F. Molecular Mechanism for Antibody-Dependent Enhancement of Coronavirus Entry. J Virol. 2020 Feb 14;94(5):e02015-19. doi: 10.1128/JVI.02015-19. Print 2020 Feb 14. PMID 31826992
- [Result] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Derived] Huang Z, Ning B, Yang HS, Youngquist BM, Niu A, Lyon CJ, Beddingfield BJ, Fears AC, Monk CH, Murrell AE, Bilton SJ, Linhuber JP, Norton EB, Dietrich ML, Yee J, Lai W, Scott JW, Yin XM, Rappaport J, Robinson JE, Saba NS, Roy CJ, Zwezdaryk KJ, Zhao Z, Hu TY. Sensitive tracking of circulating viral RNA through all stages of SARS-CoV-2 infection. J Clin Invest. 2021 Apr 1;131(7):e146031. doi: 10.1172/JCI146031. PMID 33561010